CLINICAL TRIAL: NCT00005256
Title: Coronary Screening in a High Risk Subset
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1138; R01HL043277 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-04

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

SUMMARY:
To test the hypothesis that the incidence of coronary heart disease and cardiovascular mortality could be accurately predicted by the presence of coronary calcific deposits detected by cardiac fluoroscopy.

DETAILED DESCRIPTION:
BACKGROUND:

Because of its low cost and non-invasive nature, fluoroscopy was thought to be a potentially powerful screening tool for coronary heart disease if its efficiency could be demonstrated. The utility of exercise testing for screening had been limited by its relatively low sensitivity since it could only detect atherosclerotic plaque large enough to significantly impede coronary flow.

DESIGN NARRATIVE:

Asymptomatic high risk subjects were screened with cardiac fluoroscopy and exercise testing at baseline and followed for six years with annual visits. The sensitivity and specificity of fluoroscopy in relation to the incidence of coronary heart disease and the incidence of cardiovascular mortality was determined and compared at 3.5 and 6 years of follow-up. The predictive utility of fluoroscopy and exercise testing, in relation to the incidence of coronary events, was assessed by logistic regression analysis. Multivariate analysis was also performed on baseline risk factors.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-05; Study Completion 1996-08 (Actual)

REFERENCES:
- [Background] Detrano RC, Wong ND, French WJ, Tang W, Georgiou D, Young E, Brezden OS, Doherty T, Brundage BH. Prevalence of fluoroscopic coronary calcific deposits in high-risk asymptomatic persons. Am Heart J. 1994 Jun;127(6):1526-32. doi: 10.1016/0002-8703(94)90381-6. PMID 8197979
- [Background] Detrano RC, Wong ND, Tang W, French WJ, Georgiou D, Young E, Brezden OS, Doherty TM, Narahara KA, Brundage BH. Prognostic significance of cardiac cinefluoroscopy for coronary calcific deposits in asymptomatic high risk subjects. J Am Coll Cardiol. 1994 Aug;24(2):354-8. doi: 10.1016/0735-1097(94)90287-9. PMID 8034867
- [Background] Doherty TM, Tang W, Dascalos S, Watson KE, Demer LL, Shavelle RM, Detrano RC. Ethnic origin and serum levels of 1alpha,25-dihydroxyvitamin D3 are independent predictors of coronary calcium mass measured by electron-beam computed tomography. Circulation. 1997 Sep 2;96(5):1477-81. doi: 10.1161/01.cir.96.5.1477. PMID 9315534
- [Background] Secci A, Wong N, Tang W, Wang S, Doherty T, Detrano R. Electron beam computed tomographic coronary calcium as a predictor of coronary events: comparison of two protocols. Circulation. 1997 Aug 19;96(4):1122-9. doi: 10.1161/01.cir.96.4.1122. PMID 9286939
- [Background] Detrano RC, Wong ND, Doherty TM, Shavelle R. Prognostic significance of coronary calcific deposits in asymptomatic high-risk subjects. Am J Med. 1997 Apr;102(4):344-9. doi: 10.1016/s0002-9343(97)00085-5. PMID 9217615